CLINICAL TRIAL: NCT06921798
Title: Remote Resilience: Novel Applications of mHealth in Nicaragua's Cancer Control Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Emma McKim Mitchell, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSR231558
Record Dates: First submitted 2025-02-05; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: HPV Infection; Cervical Cancers
Keywords: mHealth; Nicaragua; Cervical Cancer Screening; HPV; HPV Screening; HPV Testing
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receives cervical screening, does not receive the mHealth intervention
- Intervention (Experimental): Receives cervical screening, receives the mHealth intervention
  Interventions: Other: mHealth

INTERVENTIONS:
Other: mHealth — This mHealth intervention is designed to provide health education, and to notify study participants when their result is ready and it is time for them to return to the healthcare clinic for follow up.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test an mHealth intervention for cervical cancer prevention in under-screened women ages 25-64 on the Caribbean Coast of Nicaragua. The mHealth intervention combines a patient-centered mobile app, a provider portal, and connectivity to the National Breast and Cervical Cancer Surveillance System (SIVIPCAN). The mHealth intervention will be combined with HPV primary screening for cervical cancer. The main questions it aims to answer are, when integrated into an HPV-based screening program:

Is the mHealth intervention acceptable? Is the mHealth intervention feasible?

Researchers will compare the intervention group (mHealth intervention) to the control group (standard care).

Participants will:

Receive HPV-based cervical screening. Intervention group: Through the patient-centered app, participants will receive "results ready" notification and navigation to the clinic for follow-up.

Control group: Participants will receive "results ready" notification and navigation to the clinic for follow-up through existing communication channels.

DETAILED DESCRIPTION:
Cervical cancer, a preventable cancer of disparities, is the primary cause of cancer death for women in Nicaragua. The World Health Organization (WHO) adopted an elimination strategy for cervical cancer within the next 100 years, and outlined specific targets to meet by 2030: vaccination (90% of girls before age 15); screening/early detection (70% of women get a high-quality screen by 35 and again at 45); and treatment (90% of pre-cancerous and cancerous lesions treated). As the majority of the burden of cervical cancer exists in low- and middle-income countries (LMICs), significant research into the development, implementation, and cost-effectiveness of community-based cervical cancer screening models using HPV primary screening has developed a strong evidence-base for the acceptability and feasibility of this modality. However, significant geographic variability exists in successfully improving patient health outcomes and preventing cervical cancer, particularly in rural and remote geographic areas. In Nicaragua, significant intra-country variability exists in terms of yearly participation in cervical cancer screening by eligible women, and likelihood of lifetime screening, depending on geographic region. There is a demonstrated need for culturally tailored, regionally specific innovations in evidence-based HPV primary cervical screening programs. Researchers at the University of Virginia have worked with community partner non-governmental organization Fundacion Movicancer over the past several years to develop and create an mHealth platform that combines: (1) a patient-centered mobile application (app) called "Azulado" with (2) a provider-focused portal, as well as integration of the provider-focused portal with the (3) National Cervical Cancer Surveillance System (SIVIPCAN).

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 25-64
* Owns smart phone with Android operating system
* Lives on the Caribbean Coast of Nicaragua

Exclusion Criteria:

* Pap test or cervical screen in the last year
* Pregnant currently

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Anyone with a cervix is eligible to participate
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability/feasibility of integrating provider mHealth intervention into cervical cancer screening program | 2-4 weeks after enrollment in the study
  The Systems Usability Scale (minimum 1, maximum 5, higher scores mean more positive outcome).
Acceptability/feasibility of integrating provider mHealth intervention into cervical cancer screening program | 2-4 weeks after enrollment in the study
  (2) the uMobile App Rating Scale (minimum 1, maximum 4, higher scores mean more positive outcome).

SECONDARY OUTCOMES:
mHealth Intervention Impacts | 2-4 weeks after enrollment in the study
  1. Lost to follow-up (total number in control and intervention group)
  2. Time from initial screen through follow up treatment (measured in days)

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Mitchell, PhD, RN, Principal Investigator — University of Virginia School of Nursing

REFERENCES:
- [Background] Capote Negrin LG. Epidemiology of cervical cancer in Latin America. Ecancermedicalscience. 2015 Oct 8;9:577. doi: 10.3332/ecancer.2015.577. eCollection 2015. PMID 26557875
- [Background] Holme F, Maldonado F, Martinez-Granera OB, Rodriguez JM, Almendarez J, Slavkovsky R, Bansil P, Thomson KA, Jeronimo J, de Sanjose S. HPV-based cervical cancer screening in Nicaragua: from testing to treatment. BMC Public Health. 2020 Apr 15;20(1):495. doi: 10.1186/s12889-020-08601-z. PMID 32295562
- [Background] Mitchell EM, Lothamer H, Garcia C, Marais AD, Camacho F, Poulter M, Bullock L, Smith JS. Acceptability and Feasibility of Community-Based, Lay Navigator-Facilitated At-Home Self-Collection for Human Papillomavirus Testing in Underscreened Women. J Womens Health (Larchmt). 2020 Apr;29(4):596-602. doi: 10.1089/jwh.2018.7575. Epub 2019 Sep 18. PMID 31532298
- [Background] Mitchell EM, Hall KM, Doede A, Rong A, McLean Estrada M, Granera OB, Maldonado F, Al Kallas H, Bravo-Rodriguez C, Forero M, Pokam Tchuisseu Y, Dillingham RA. Feasibility and acceptability of self-collection of Human Papillomavirus samples for primary cervical cancer screening on the Caribbean Coast of Nicaragua: A mixed-methods study. Front Oncol. 2023 Jan 20;12:1020205. doi: 10.3389/fonc.2022.1020205. eCollection 2022. PMID 36741739